CLINICAL TRIAL: NCT02712281
Title: Autism MEAL Plan: Parent Training to Manage Eating Aversions & Limited Variety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, William Sharp, PhD, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00085811
Record Dates: First submitted 2016-03-09; First posted 2016-03-18 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Food Selectivity; Autism MEAL Plan; Parent Education
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autism MEAL Plan (Experimental): Parents of eligible children who are randomized to the Autism Managing Eating Aversions and Limited variety (MEAL) Plan will participate in group-based parent training sessions (4 parents per group).
  Interventions: Behavioral: Autism MEAL Plan
- Parent Education (Active Comparator): Parents of eligible children who are randomized to the Parent Education Arm will receive group-based parent education (PE). Each group includes 4 parents.
  Interventions: Behavioral: Parent Education

INTERVENTIONS:
Behavioral: Autism MEAL Plan — The Autism MEAL plan includes education on feeding issues and behavior management, and specific strategies to expand dietary diversity. Each parent receives 1.5 hours of intervention per week for 10 weeks by a masters or doctoral level clinician. The first three sessions focus on understanding feeding problems and behavior management strategies in children with ASD.The next seven sessions include child-specific feeding interventions, based on parent-report and home data collection of child meal time behavior. To promote application of new skills, homework accompanies each lesson.
  The next seven sessions include child-specific feeding interventions, based on parent-report and home data collection of child meal time behavior. To promote application of new skills, homework accompanies each lesson.
  Arms: Autism MEAL Plan
Behavioral: Parent Education — The Parent Education study arm includes 10 sessions focusing on the following topics: understanding Autism Spectrum Disorder (ASD), clinical assessments for ASD, development in children with ASD, medical and genetic comorbidities in ASD, family and sibling issues, treatment alternatives, and education and treatment planning. The Parent Education arm does not include topics related to feeding problems or feeding specific interventions. Each parent receives 1.5 hours of intervention per week for 10 weeks by a masters or doctoral level clinician.
  Children randomized to Parent Education will be offered the Autism MEAL Plan after completing the 10-week randomized trial.
  Arms: Parent Education

SUMMARY:
The Autism Managing Eating Aversions and Limited variety (MEAL) Plan is a group-based parent training intervention designed to assist parents in increasing the variety of foods eaten in children with Autism Spectrum Disorder (ASD). The goal of the Autism MEAL Plan is to include specific techniques to manage mealtime behavioral challenges and introduce new foods.

DETAILED DESCRIPTION:
The Autism Managing Eating Aversions and Limited variety (MEAL) Plan is a structured parent-mediated, group-based intervention to reduce mealtime disruptive behavior, expand dietary diversity and reduce parental stress associated with moderate food selectivity in young children with Autism Spectrum Disorder (ASD).

Children ages 3-8 with a diagnosis of ASD who present with moderate food selectivity and associated problem behavior will be screened for inclusion in the study. Following consent and screening procedures, parents of eligible children will be assigned to a group-based parent training (Autism MEAL plan) or group-based parent education. Each parent will receive 1.5 hours of intervention per week for 10 weeks by a masters or doctoral level clinician.

Data will be collected on parental compliance with the Autism MEAL plan and the food acceptance of the child as well as nutritional intake, and refusal behaviors. Child participants will also be included in parent-child dyad in-vivo feedback sessions. Parents assigned to parent education will be able to cross-over to receive the Autism MEAL Plan following completion of post-study measures.

The first aim of the study is to finalize the Autism MEAL Plan materials (e.g., role-play activities, activity sheets and video examples). This includes standardizing therapist scripts in line with the revised curriculum and creating new video examples that coincide with practice worksheets. Home recording (e.g., personal camera phone) to document and present home meal data will also be added to the curriculum.

The second aim is to evaluate the feasibility of the Autism MEAL Plan versus parent education in 40 children (20 per treatment assignment) with ASD and moderate feeding problems.

The final study aim is to evaluate the preliminary efficacy of the Autism MEAL Plan in expanding food diversity, decreasing disruptive behavior and reducing parental stress compared to Parent Education. Methods of evaluating this aim include direct observation, parent ratings of behavior, food intake and stress, as well as blinded clinician ratings, height, weight and BMI.

ELIGIBILITY:
Inclusion Criteria (for children):

* A diagnosis of autism spectrum disorder (ASD), supported by the Autism Diagnostic Observation Schedule (ADOS) and the Social Communication Questionnaire (SCQ)-Lifetime
* Presents with a history of moderate food selectivity (a diet involving at least 6 food items)
* Accepting at least one fruit or vegetable
* Fewer than two food items in one or more food categories (i.e., fruit, vegetable, protein, starch) as measured by the Food Preference Inventory
* Exhibits disruptive refusal behaviors when presented with non-preferred foods (e.g., crying, active verbal protest, tantrums) often or during every meal as indicated by item 7 on the Brief Autism Mealtime Behavior Inventory (BAMBI)

Inclusion Criteria (for parents or primary caregivers):

* Parent, or primary caregiver, endorses a feeding concern as one of the top two problems on the Parent Target Problem
* Parent, or primary caregiver, agrees to participate and is deemed able to attend group sessions
* Parent, or primary caregiver, is able to speak, understand, read and write in English

Exclusion Criteria (for children):

* Severe feeding problems (e.g., < 5 preferred foods as measure by the Food Preference Inventory)
* Complex medical issues (e.g., gastrostomy tube or formula dependent) requiring intensive treatment such as day treatment or hospital-based treatment

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2016-07; Primary Completion 2018-03 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Global Impression - Improvement scale (CGI-I) score | Baseline, end of follow-up (up to 18 weeks)
  The Clinical Global Impression - Improvement scale (CGI-I) is a 7-point scale measure of overall change of Parent Target Problems (the child's two most pressing problems at screening, as reported by parents), using scores from the Clinical Global Impressions - Severity scale (CGI-S). Scores range from 1 (Very Much Improved) through 4 (Unchanged) to 7 (Very Much Worse).

SECONDARY OUTCOMES:
Change in Parenting Stress Index- Short Form (PSI) score | Baseline, end of follow-up (up to 18 weeks)
  The Parenting Stress Index- Short Form (PSI) is a 36-item survey commonly used
Parent Satisfaction Rating | Week 14
  A 10 item Parent Satisfaction Rating questionnaire will assess acceptance and perceived effectiveness of each treatment arm.
Change in Brief Autism Mealtime Behavior Inventory (BAMBI) scores | Baseline, end of follow-up (up to 18 weeks)
  The Brief Autism Mealtime Behavior Inventory (BAMBI) is an 18-item parent-rated questionnaire on mealtime behaviors
Change in Food Preference Inventory (FPI) scores | Baseline, end of follow-up (up to 18 weeks)
  A 154-item parent-rating of food selectivity. It includes seven food categories (fruits, vegetables, proteins, starches, dairy, miscellaneous/snack, combination foods. The food selectivity score = the number of foods reported as "never" consumed divided by 154 X 100. We will also derive a food acceptance score = the number of food items endorsed as accepted divided by 154 X 100.
Change in nutritional intake | Baseline, end of follow-up (up to 18 weeks)
  Nutritional intake will be assessed by parents recording the child's daily intake on a food diary for 3 days prior to the Baseline, Week 10, Week 14, and Week 18 visits. A nutritionist (blind to treatment assignment) will tally the child's intake of selected vitamins and nutrients (vitamins A, C, D, and E, zinc, calcium, iron, fiber, fat, protein, carbohydrates, and total energy [kcal]) to determine the overall level of each micro- and macro-nutrient. The total number of nutrient deficiencies will be determined using cut points. The evaluation of change in nutritional status will be assessed by averaging the levels of each nutrient across groups.
Change in Aberrant Behavior Checklist (ABC) scores | Baseline, end of follow-up (up to 18 weeks)
  The Aberrant Behavior Checklist (ABC) is a commonly used 58-item parent-rated measure of overall behavioral problems. Subscale categories of the ABC include: Irritability, Lethargy, Stereotypy, Hyperactivity, and Inappropriate Speech.
Change in rapid acceptance during 10 minute meal observation | Baseline, end of follow-up (up to 18 weeks)
  Children and parents will participate in a 10-minute meal observation at the Baseline, Week 10, Week 14 and Week 18 visits. During the 10-minute meal observation caregivers are instructed to present a small bite of food to the child at 30-second intervals with a preset group of foods (e.g., green beans, peaches, grilled chicken, potatoes). Data are collected on a variety of mealtime behaviors including rapid acceptance of food presented. Outcomes are rated by trained observers using conventions established in the Marcus Autism Center's Feeding Disorders Program.
Change in rapid swallowing during 10-minute meal observation | Baseline, end of follow-up (up to 18 weeks)
  Children and parents will participate in a 10-minute meal observation at the Baseline, Week 10, Week 14 and Week 18 visits. During the 10-minute meal observation caregivers are instructed to present a small bite of food to the child at 30-second intervals with a preset group of foods (e.g., green beans, peaches, grilled chicken, potatoes). Data are collected on a variety of mealtime behaviors including rapid swallowing of food presented. Outcomes are rated by trained observers using conventions established in the Marcus Autism Center's Feeding Disorders Program.
Change in disruptions during 10-minute meal observation | Baseline, end of follow-up (up to 18 weeks)
  Children and parents will participate in a 10-minute meal observation at the Baseline, Week 10, Week 14 and Week 18 visits. During the 10-minute meal observation caregivers are instructed to present a small bite of food to the child at 30-second intervals with a preset group of foods (e.g., green beans, peaches, grilled chicken, potatoes). Data are collected on a variety of mealtime behaviors including disruptions (e.g. head turning, pushing away the spoon) when food is presented. Outcomes are rated by trained observers using conventions established in the Marcus Autism Center's Feeding Disorders Program.
Change in crying during 10-minute meal observation | Baseline, end of follow-up (up to 18 weeks)
  children and parents will participate in a 10-minute meal observation at the Baseline, Week 10, Week 14 and Week 18 visits. During the 10-minute meal observation caregivers are instructed to present a small bite of food to the child at 30-second intervals with a preset group of foods (e.g., green beans, peaches, grilled chicken, potatoes). Data are collected on a variety of mealtime behaviors including crying when food is presented. Outcomes are rated by trained observers using conventions established in the Marcus Autism Center's Feeding Disorders Program.
Change in volume of food consumed during 10-minute meal observation | Baseline, end of follow-up (up to 18 weeks)
  Children and parents will participate in a 10-minute meal observation at the Baseline, Week 10, Week 14 and Week 18 visits. During the 10-minute meal observation caregivers are instructed to present a small bite of food to the child at 30-second intervals with a preset group of foods (e.g., green beans, peaches, grilled chicken, potatoes). The volume of food consumed will be measured to assess changes in intake. Outcomes are rated by trained observers using conventions established in the Marcus Autism Center's Feeding Disorders Program.
Weight | Baseline, end of follow-up (up to 18 weeks)
  Direct measurement of weight using a digital scale recorded in kg.
Height | Baseline, end of follow-up (up to 18 weeks)
  Direct measurement of height using a stadiometer recorded in cm.
Body Mass Index | Baseline, end of follow-up (up to 18 weeks)
  Height and weight measurements will be used to calculate BMI percentile by age for each participant and converted to age- and sex- adjusted Z-scores based on the 2000 CDC growth charts

CONTACTS AND LOCATIONS:
Overall Officials: William Sharp, PhD, Principal Investigator — Emory University
Locations (1):
- Marcus Autism Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharp WG, Burrell TL, Berry RC, Stubbs KH, McCracken CE, Gillespie SE, Scahill L. The Autism Managing Eating Aversions and Limited Variety Plan vs Parent Education: A Randomized Clinical Trial. J Pediatr. 2019 Aug;211:185-192.e1. doi: 10.1016/j.jpeds.2019.03.046. Epub 2019 May 3. PMID 31056202